CLINICAL TRIAL: NCT04032015
Title: Randomized, Sham-controlled rTMS Trial in Depression to Evaluate the Relationship of Brain Plasticity and Clinical Outcome
Brief Title: rTMS Study in Depression to Evaluate the Relationship Between Brain Plasticity and Clinical Outcome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not currently active
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Corey Keller, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 133611
Record Dates: First submitted 2019-07-22; First posted 2019-07-25 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- rTMS treatment (Active Comparator): rTMS will be delivered for 20 sessions over 4 weeks. Active 10 Hz rTMS will be delivered using neuro-navigation based on participants' own MRI images. Daily treatment regiments will last 30 minutes and rTMS will be delivered at 120% of the participant's motor threshold. Participants will be monitored during the rTMS sessions for adverse events and/or side effects.
  Interventions: Device: TMS
- Sham treatment (Sham Comparator): Sham rTMS will be delivered for 20 sessions over 4 weeks. To maximize sham validity, both 1) a direction-sensor TMS coil will alert the operators to flip the coil if the wrong side is being used, and 2) low-intensity 10Hz electrical stimulation will be applied to scalp electrodes under the coil for sham and placed but not activated in the active arm. The rTMS coil will be positioned using neuro-navigation based on participants' own MRI images, mimicking active rTMS treatment. Daily treatment regiments will last 30 minutes and sham rTMS will be delivered at 120% of the participant's motor threshold. Participants will be monitored during the sham rTMS sessions for adverse events and/or side effects.
  Upon completing the 20 sham sessions, participants are unblinded and offered 20 treatments of active rTMS. The open-label treatment would follow the active rTMS treatment protocol.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Device used to administer electromagnetic fields to the brain to alter connectivity patterns

SUMMARY:
Depression is a highly prevalent condition characterized by persistent low mood, energy, and activity that can affect one's thoughts, mood, behavior, and sense of well-being. Repetitive transcranial magnetic stimulation (rTMS), a non-invasive neuromodulatory technique, is an effective treatment for depression. However, remission rates are suboptimal and ideal stimulation parameters are unknown. The overarching goal of this study is to elucidate how brain changes accumulate during rTMS, and how these changes relate to clinical outcome. I plan to recruit patients with medication-resistant depression and treat with four weeks of rTMS in a randomized, double-blind, sham-controlled fashion. I will measure brain changes using TMS-EEG and determine how these changes relate to clinical outcome. This study will 1) test how brain changes relate to clinical outcome and 2) establish a computational model to help predict outcome and propose novel treatment protocols.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an effective treatment for major depressive disorder, but remission rates are 20-40%, and ideal stimulation parameters are unknown. rTMS is thought to work by changing the synaptic strength of neurons. The ability of our brain to make these changes is referred to as plasticity. rTMS-induced changes are thought to build with successive treatment sessions, a process referred to as metaplasticity. While both plasticity and metaplasticity are well-established in single cell physiology, relevance to rTMS in humans remains unknown. To improve clinical efficacy, the investigators seek to understand 1) the neural response to a single rTMS session (plasticity), 2) the neural response to repeated daily rTMS sessions (metaplasticity), and 3) whether computational models of plasticity based on single-cell physiology apply to human patients receiving rTMS for depression.

Goals of the study are as follows:

1. establish a detailed mechanistic understanding of the brain changes during current rTMS treatment
2. identify clinically meaningful electrophysiological biomarkers for rTMS treatment
3. establish a computational model to help predict both brain and clinical changes.

This project tests the hypothesis that neural changes that accumulate during rTMS treatment can predict clinical outcome. Participants will first complete a screening procedure to determine eligibility based on the inclusion/exclusion criteria. If the participants are not eligible, no further study procedures will be conducted. Eligible participants will be randomized to four weeks (20 sessions) of daily 10Hz left dorsolateral prefrontal cortex (DLPFC) active or sham rTMS. Following the completion of sham treatment, participants will be offered open-label active rTMS treatment for four weeks to ensure that all participants receive active treatment if desired. Single pulse TMS-evoked potential (TEP), a well-studied causal EEG measure of brain excitability, will be measured before, during, and after every rTMS session. TEPs will be measured locally in the left lateral prefrontal cortex and compared to downstream sites in parietal and medial prefrontal cortex.

Aim 1: To determine the electrophysiological response to single and repeated rTMS sessions in depression. Through this aim, I will establish a detailed mechanistic understanding of the electrophysiological effects of rTMS treatments.

Aim 2: To determine the relationship between brain state, plasticity, metaplasticity, and antidepressant response in depression. Through this aim, I will identify clinically meaningful electrophysiological biomarkers for rTMS treatment.

Aim 3: To test whether a computational model of metaplasticity applies to human patients. This computational model will help predict both neurophysiological and clinical changes.

Findings from this study will provide the basis for novel stimulation protocols that will maximize clinically-relevant brain changes and improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Right-handed
* Ages 18-65
* Depression diagnosis as assessed through an in-depth interview
* Failed at least 1 antidepressant medication
* Without current/history of neurological disorders or seizures or risk of seizures

Exclusion Criteria:

* A contraindication for MRIs (e.g. implanted metal)
* History of head trauma with loss of consciousness
* History of seizures
* Neurological or uncontrolled medical disease
* Active substance abuse
* Diagnosis of psychotic or bipolar disorder
* Prior history of ECT or rTMS failure
* Currently taking medications that substantially reduce seizure threshold
* Currently pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
TMS-EEG change | Up to 1 month
  Change in TMS-EEG measures will be assessed before, during, and after each treatment session. These changes will be compared to clinical outcome to identify clinically-relevant biomarkers.
Hamilton Depression Rating Scale (HamD) | Up to 6 months after treatment
  Clinician administered scale to assess depression is a 24-item clinician-administered assessment utilized as a way of determining a patient's level of depression before, during, and after treatment. It takes approximately 15-20 minutes to complete the interview and score the results.

IPD SHARING:
Plan to Share IPD: Undecided